CLINICAL TRIAL: NCT07175805
Title: Pelvic Floor Disorder Symptoms in Women Seeking Weight Loss Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Hartford HealthCare (Other)
Responsible Party: Principal Investigator, Madeline Carmain, Fellow, Urogynecology, Hartford HealthCare
Other Study IDs: HHC-2025-0168
Record Dates: First submitted 2025-07-28; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Lower Urinary Tract Symptoms; Stress Urinary Incontinence; Urge Urinary Incontinence; Overactive Bladder; Pelvic Organ Prolapse; Weight Loss; Fecal Incontinence; Bariatric Surgery; glp1 Agonist
Keywords: lower urinary tract symtpoms; stress urinary incontinence; urge urinary incontinence; overactive bladder; pelvic organ prolapse; weight loss; fecal incontinence; bariatric surgery; glp1 agonist
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Bladder, Overactive; Pelvic Organ Prolapse; Weight Loss; Fecal Incontinence | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bariatric Surgery: Patients who plan to undergo bariatric surgery
  Interventions: Procedure: Bariatric Surgery
- GLP1 or GLP1/GIP1: Patients who plan to take GLP1 or GLP1/GIP1 medications
  Interventions: Drug: GLP1 receptor agonist

INTERVENTIONS:
Procedure: Bariatric Surgery — Patients in this arm plan to undergo gastric sleeve or gastric bypass surgery.
  Groups: Bariatric Surgery
Drug: GLP1 receptor agonist — Patients in this arm plan to start a GLP-1 receptor agonist.
  Groups: GLP1 or GLP1/GIP1

SUMMARY:
The purpose of this study is to compare change in pelvic floor symptoms between patients receiving medical therapy for weight loss and surgical treatment for weight loss. Examples of pelvic floor symptoms include urinary incontinence, urinary urgency, urinary frequency, fecal incontinence, and vaginal prolapse. Participants in this study do not need to have any pelvic floor symptoms to enroll in the study. Understanding how different types of weight loss treatment impact pelvic floor symptoms will help clinicians guide which weight loss treatments are recommended for patients with pelvic floor symptoms in the future.

DETAILED DESCRIPTION:
Lower Urinary Tract Symptoms (LUTS) are defined as bothersome symptoms related to the storage of urine, voiding, and postvoid symptoms, and includes urgency, frequency, and urinary incontinence (UI). UI is the involuntary loss of urine and is a common and bothersome form of LUTS. The prevalence of urinary incontinence is high and increasing, with 61.8% of all women over 20 years old reporting urinary incontinence. High body mass index (BMI) is associated with higher risk of UI. In women with UI, modest weight loss due to behavioral changes or dieting has been shown to decrease the frequency of UI episodes. In women with UI who lost weight through bariatric surgery, there is improvement or even complete resolution of UI symptoms. Within the field of weight loss management, bariatric surgery is seen as the gold standard treatment with well-established improvements in LUTS symptoms.

UI is known to impact quality of life, with worse UI symptoms correlated with worse quality of life scores. Treatment resulting in improved or resolution of UI symptoms improves quality of life scores. In addition, UI takes a financial toll on women, with estimates from 2008 showing that patients spend $1500 annually for incontinence products. Any treatment which is able to improve or resolve symptoms of UI has the potential to significantly improve patient's quality of life and decrease patient's financial burdens.

In addition to LUTS symptoms, there are other pelvic disorders which are influenced by obesity and pelvic muscle function. Pelvic organ prolapse (POP), the descent of intrabdominal organs (bladder, rectum, intestines, uterus) into the vaginal space, is more common in overweight and obese women; a metanalysis of women with POP who underwent bariatric surgery had improvement in POP symptoms after surgery. Fecal incontinence (FI) is the involuntary loss of stool; the rate of FI is higher in patients with obesity. The causal relationship between weight loss and FI improvement is not clear (as FI is highly dependent on stool consistency), although there are studies which demonstrate improvement of FI after bariatric surgery. All of these disorders can be treated or improved with pelvic floor physical therapy, illustrating the importance of pelvic floor musculature in appropriate function of pelvic organs and function. A weight loss therapy which potentially diminishes the function of the pelvic floor through lean muscle loss may worsen any of these pelvic floor associated disorders.

In 2021, semaglutide, a glucagon-like peptide-1 receptor agonist (GLP-1 RA), was approved by the FDA for weight management. Since this approval, there has been a rapid uptake of these medications for weight loss, with 1 in 12 people in the United States having been prescribed a GLP-1 RA as of May 2024. A recent study showed that GLP-1 RA prescriptions for people who were overweight or obese but did not have diabetes increased 700% between 2019 and 2023. With the rapid uptake of these drugs for weight loss, there has been significant interest in understanding the full beneficial effects of treatment for patients taking GLP-1 RA for weight loss, with recent studies demonstrating cardiovascular benefits for overweight patients being treated with GLP-1 RAs. A second class of related medications, dual GLP-1 RA and gastric inhibitory peptide-1 (GIP1) medications have been released and are being used for weight loss management. At this time, there are no studies published investigating the effect of weight loss with GLP-1 RAs or GLP-1/GIP1s on LUTS.

Given the rapid uptake of this therapy class for weight loss, it is necessary to establish whether weight loss from GLP-1 RAs results in the same improvement in LUTS as other therapies. Recent investigations show that there can be a high amount of lean body mass and muscle loss as a component of the weight lost with GLP-1 RA therapy; recent studies demonstrate that 30% of weight lost using GLP-1 RAs was secondary to loss of lean muscle mass. As the pelvic floor musculature is essential in preventing LUTS symptoms, GLP-1 RA therapy may worsen LUTS. At this time, it is not clear that weight lost with GLP-1 RAs will result in the same improvement of LUTS symptoms as weight lost with behavioral changes, dietary changes, or bariatric surgery.

In this study, the investigators will evaluate the difference of LUTS, UI, FI, and POP symptoms between patients losing weight through bariatric surgery or GLP-1/GIP1 therapy. By comparing results of weight loss from GLP-1 RAs or combination GLP-1/GIP1 medications to weight loss from bariatric surgery, the gold standard weight loss treatment that is well established to improve LUTS and POP symptoms, the investigators will be able to detect whether there are differences in improvement in these pelvic floor disorders based on the mechanism of weight loss or whether it is only the amount of weight lost that impacts symptomatic improvement.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18-89 years old
* any race/ethnicity
* BMI ≥30 kg/m2
* current medical weight loss or surgical weight loss patient of Obesity Medicine and Metabolic & Bariatric Surgery
* able/willing to give informed consent
* have a home scale to measure weight

Patients meeting all the following criteria will be eligible to participate in the medical weight loss therapy arm:

* prescribed and start a glucagon-like peptide-1 receptor agonist (GLP-1 RA) or a GLP-1/gastric inhibitory peptide (GIP1)
* taking other weight loss agents (such as metformin)

Patients meeting all the following criteria will be eligible to participate in the bariatric surgery arm:

* plan to undergo gastric sleeve or gastric bypass surgery
* taking weight loss agents which are not GLP-1 RA or GLP-1/GIP1 medications at the start of the study. Patients will not be excluded if they are started on GLP-1 RA or GLP-1/GIP1 medications after surgery.

Exclusion Criteria:

* Pregnant
* ≥90 years old
* <18 years old
* BMI <30 kg/m2
* A history of bariatric surgery prior to enrollment
* No home scale to measure weight
* Active cancer

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seeking medical weight loss or surgical weight loss at the weight loss clinics at Hartford Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in pelvic floor symptoms measured by survey the Urogenital Distress Inventory (UDI) | 6 months
  The investigators plan to measure the change in pelvic floor symptoms between woman taking glucagon-like peptide-1 receptor agonists (GLP1) medications vs women receiving bariatric surgery. These changes will be measured by validated survey, including the Urogenital Distress Inventory (UDI)
Change in pelvic floor symptoms measured by validated survey the Colorectal-Anal Distress Inventory (CRADI-8). | 6 months
  The investigators plan to measure the change in pelvic floor symptoms between woman taking glucagon-like peptide-1 receptor agonists (GLP1) medications vs women receiving bariatric surgery. These changes will be measured by validated survey the Colorectal-Anal Distress Inventory (CRADI-8).

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No